CLINICAL TRIAL: NCT04812782
Title: Influence Of Extra Virgin Olive Oil and Butter on Endothelial Function in Type 1 Diabetes
Brief Title: Dietary Fat and Endothelial Function in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Concetta Irace, Clinical Professor, University Magna Graecia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Dietary Fat in Type 1 Diabetes
Record Dates: First submitted 2021-03-12; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Type 1 Diabetes
Keywords: Endothelial function; FMD; gastric emptying; post prandial glycemia; dietary fat; EVOO; butter
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Cross-over, interventional, controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVOO-Butter (Experimental): All patients and control subjects who met inclusion and exclusion criteria, and signed the Informed Consent, were scheduled for the two study visits, one week apart, during which each participant received two types of high GI meal: the first enriched with EVOO and the second with butter.
  Interventions: Dietary Supplement: EVOO supplementation; Dietary Supplement: Butter supplementation
- Butter-EVOO (Experimental): All patients and control subjects who met inclusion and exclusion criteria, and signed the Informed Consent, were scheduled for the two study visits, one week apart, during which each participant received two types of high GI meal: the first enriched with Butter and the second with EVOO
  Interventions: Dietary Supplement: EVOO supplementation; Dietary Supplement: Butter supplementation

INTERVENTIONS:
Dietary Supplement: EVOO supplementation — We will administer to both groups (healthy and T1D subjects) a high glycemic index meal enriched with EVOO
Dietary Supplement: Butter supplementation — We will administer to both groups (healthy and T1D subjects) a high glycemic index meal enriched with butter

SUMMARY:
The purpose of this study is to evaluate the effects of the add-on of extra vergin olive oil or butter to a high glycemic index meal on endothelial function in subjects with type 1 Diabetes and healthy subjects.

DETAILED DESCRIPTION:
Impaired endothelial function is an early manifestation of atherosclerosis and predictor of incident cardiovascular events. Diabetes affects arterial vasodilation by reducing the bioavailability of NO and more in general affecting the balance between the atheroprotective and atherothrombotic properties of the endothelium. A consistent number of studies has so far documented that Mediterranean-style diet associates with reduced risk of cardiovascular diseases and diabetes. Intake of extra virgin olive oil (EVOO), that is a common but not necessary ingredient of the Mediterranean diet, seems to further enhance the beneficial cardiovascular effect and reduce the incidence of diabetes. We have designed the present study to test whether EVOO supplementation acutely influences endothelial function in T1DM. EVOO supplementation wil be compared to butter supplementation in the context of a high glycemic index (GI) meal that is known to increase PP glycemic burden.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years,
* diagnosis of type 1 diabetes since at least 1 year,
* HbA1c <8.5% (69 mmol/mol),
* stable insulin therapy for at least 3 months before the enrolment into the study

Exclusion Criteria:

* pregnancy, celiac disease, history of cardiovascular diseases, hypertension, hyperlipidemia, retinopathy, nephropathy, neuropathy, and ongoing treatment with vasoactive drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Change of Endothelial function from pre meal to post meal period | before meal, 1 hour, 3 hour, 5 hour after meal
  Flow mediated dilation technique by ultrasound

SECONDARY OUTCOMES:
Serum glucose | before meal, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour after meal
  glucose-hexokinase method
Gastric emptying rate | before meal, 15, 90, 120, 180, 240, 300 minutes after meal
  Ultrasound antrum measurement

CONTACTS AND LOCATIONS:
Locations (1):
- University Magna Graecia, Catanzaro, Italy